CLINICAL TRIAL: NCT01370330
Title: 131I-Labeled MIBG for Refractory Neuroblastoma: A Compassionate Use Protocol
Status: Available | Type: Expanded Access
Sponsor: Kieuhoa Vo (Other)
Collaborators: Cannonball Kids' Cancer Foundation (Other)
Responsible Party: Sponsor-Investigator, Kieuhoa Vo, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Other Study IDs: CompUse MIBG; NCI-2011-01902 (Registry Identifier: NCI Clinical Trials Reporting Program); 05161 (Other: University of California, San Francisco)
Record Dates: First submitted 2011-05-27; First posted 2011-06-09 (Estimated); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; MIBG; 131I-MIBG; Resistant; Relapsed; Treatment; University of California, San Francisco; Pediatric; Oncology
MeSH Terms: conditions — Neuroblastoma; Recurrence; Neoplasms | interventions — 3-Iodobenzylguanidine

INTERVENTIONS:
Drug: Metaiodobenzylguanidine (MIBG) — 131I-MIBG Therapeutic Administration. Therapeutic 131I-MIBG will be synthesized at Jubilant DraxImage (Quebec, Canada) with specific activities of 9-18 Ci/mmole, or at Progenics with specific activity of 2,500 mCi/mg. The therapeutic dose (8-18 mCi/kg at investigator's discretion; any dose greater than 12 requires stored stem cells) will be diluted in 25-50 ml of normal saline for either preparation, and will be infused intravenously through a patient's central line, if already present, or a peripheral IV if a central line is not present.If Azedra is used, the dose will be infused over 30-60 minutes; the low specific activity preparation from Draximage will be infused over 90-120 minutes. For patients with pheochromocytoma or paraganglioma, the recommended maximum dose is 500 mCI or 12 mCi/kg.
  Other Names: 131I-MIBG

SUMMARY:
This is a compassionate use protocol to allow patients with advanced neuroblastoma palliative access to 131I-metaiodobenzylguanidine (131I-MIBG).

DETAILED DESCRIPTION:
Neuroblastoma remains a fatal disease for a large percentage of patients, especially those with high-risk disease features who become resistant to conventional therapy. 131I-metaiodobenzylguanidine (131I-MIBG) is a norepinephrine analog that concentrates in adrenergic tissue and therefore holds promise for cell-specific treatment of neuroblastoma. 131I-MIBG is active against relapsed or refractory neuroblastoma and associated hematopoietic toxicity can be abrogated with autologous stem cell rescue. 131I-MIBG given in doses of 10-18 millicurie (mCi)/kg with stem cell rescue, if necessary, is safe and effective palliative therapy for refractory or relapsed neuroblastoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Refractory or relapsed neuroblastoma with original diagnosis based on tumor histopathology or elevated urine catecholamines with typical tumor cells in the bone marrow. Refractory, progressive or metastatic pheochromocytoma/paraganglioma or related tumor.
* MIBG uptake: Tumors must be shown to be MIBG avid within 6 weeks prior to enrollment
* Age > 1 year and able to cooperate with radiation safety restrictions during therapy period. Patients with pheochromocytoma/paraganglioma and related tumors must be between 1 and 12 years of age.
* Life Expectancy: greater than 6 weeks.
* Lansky and Karnofsky Performance Status: 60% or higher.
* Disease status: Failure to respond to standard therapy (usually combination chemotherapy with or without radiation and surgery) or development of progressive disease at any time (any new lesion or an increase in size of >25% of a pre-existing lesion). Disease evaluable by MIBG scan must be present within 6 weeks of study entry and subsequent to any intervening therapy.
* Stem cells: Patients must have an autologous hematopoietic stem cell product available for re-infusion after MIBG treatment at doses of >12 mCi/kg if needed. The minimum quantity for purged or unpurged peripheral blood stem cells is 1.0 x 10^6 cluster of differentiation 34 (CD34)+ cells/kg (optimum > 2 x 10^6 CD34+ cells/kg). The minimum dose for bone marrow is 1.0 x 10^8 mononuclear cells/kg (optimum > 2.0 x 10^8 mononuclear cells/kg). If no stem cells are available, then the dose of 131I-MIBG should be <12 mCi/kg .
* Prior Therapy: Patients may enter this study with or without re-induction therapy for recurrent tumor. Patients must have fully recovered from the toxic effects of any prior therapy. At least 2 weeks should have elapsed since any anti-tumor therapy and the patient must meet hematologic criteria below. Three months should have elapsed in the case of completing radiation to any of the following fields: craniospinal, total abdominal, whole lung, total body irradiation). Cytokine therapy [eg granulocyte-colony stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), interleukin-6 (IL-6), erythropoietin] must be discontinued a minimum or 24 hours prior to MIBG therapy. Prior 131I-MIBG therapy is allowed if > 6 months previous and if the patient has adequate hematopoietic stem cells available and if cumulative 131I-MIBG dose will not exceed 60 mCi/kg.
* Organ Function
* Liver function: bilirubin <2x normal and aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) < 10x normal.
* Kidney function: Creatinine less than or equal to 2
* Hematopoietic Criteria Patients must have adequate hematopoietic function (without transfusion): absolute neutrophil count (ANC) >.750 x 10E9/L; Platelets >50 x 10E9/L if stem cells are not available; if stem cells are available, the patient should be independent of platelet transfusions with a platelet count of at least 20 x 10E9/L. Hemoglobin >10g/dl at time of treatment (transfusion allowed). Patients with granulocytopenia and/or thrombocytopenia due to tumor metastatic to the bone marrow may be eligible after discussion with study chair or designee.
* Normal lung function as manifested by no dyspnea at rest or exercise intolerance, no oxygen requirement.
* No clinically significant cardiac dysfunction
* Signed informed consent: The patient and/or the patient's legally authorized guardian must acknowledge in writing that consent to become a study subject has been obtained, in accordance with institutional policies approved by the U.S. Department of Health and Human Services.

Exclusion Criteria:

* Patients with disease of any major organ system that would compromise their ability to withstand therapy. Any significant organ impairment should be discussed with the Study Chair or Vice Chair prior to patient entry.
* Because of the teratogenic potential of the study medications, no patients who are pregnant or lactating will be allowed. Patients of childbearing potential must practice an effective method of birth control while participating on this study, to avoid possible pregnancy.
* Patients who are on hemodialysis.
* Patients with active infections that meet grade 3-4 toxicity criteria.
* Patients with pheochromocytoma or paraganglioma who have any proteinuria on urinalysis must have a 24-hr urine collection for protein. If there is proteinuria above the reference range on a 24-hour urine collection, they are excluded due to increased risk of respiratory complications.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Kieuhoa Vo, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States